CLINICAL TRIAL: NCT03017651
Title: An Evaluation of a Proprietary Omega-3 Fatty Acid Incorporated Into a MAG on Blood EPA and DHA Levels: a PK Study
Brief Title: An Evaluation of Omega-3 Fatty Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Miami Research Associates (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 16.20.CLI
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OM3-supplement 1 (Experimental): 1 g capsule for OM3-supplement 1 given once
  Interventions: Dietary Supplement: OM3-supplement 1
- OM3-supplement 2 (Active Comparator): 1 g capsule for OM3-supplement 2 given once
  Interventions: Dietary Supplement: OM3-supplement 2

INTERVENTIONS:
Dietary Supplement: OM3-supplement 1 — 1g of OM3-supplement 1 will be given to subjects to look at DHA/EPA blood absorption
  Arms: OM3-supplement 1
Dietary Supplement: OM3-supplement 2 — 1g of OM3-supplement 2 will be given to subjects to look at DHA/EPA blood absorption
  Arms: OM3-supplement 2

SUMMARY:
This protocol will determine the pK profile of two different omega-3 fatty acid supplements on plasma EPA and DHA levels.

DETAILED DESCRIPTION:
This protocol is to assess the omega-3 blood levels of DHA and EPA following a single dose administration of study products by means of pharmacokinetics over a 24 hour period of time (post-dose).

ELIGIBILITY:
Inclusion criteria:

1. Male or female subjects between 18 and 65 years old (inclusive)
2. Body Mass Index (BMI) between 25.0 and 34.9 kg/m2 (inclusive) at Screening.
3. Subjects with normal or moderately elevated lipidemia (borderline lipids as defined by the AACE - Total cholesterol ≤ 240 mg/dl; LDL ≤ 160 mg/dl; TG ≤ 199 mg/dl).
4. Subjects with no clinically significant findings in the physical examination, medical history, vital signs, clinical laboratory test (hematology and serum chemistry) results and as deemed by the Investigator.
5. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign the informed consent indicating voluntary consent to participate in the study prior to the initiation of Screening or study related activities.
6. Male and female subjects of childbearing potential must agree to use one of the following medically acceptable contraceptive methods for the duration of the study: same-sex partner; double barrier (condom, diaphragm or cervical cap with spermicidal foam, gel or cream); IUD (with or without hormones) in place or hormonal contraception (oral, injectable, implantable, transdermal or vaginal) used consecutively for at least 3 months prior to study product administration; vasectomized partner or sterilization by bilateral insertion of Essure® or similar product for 6 months minimum prior to study product administration; bilateral tubal ligation, hysterectomy and/or bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to study product administration

Exclusion Criteria:

1. Currently using fish oil capsules (supplements or prescription products).
2. Regular use of omega-3 supplements (defined as greater than 500 mg/week) within 4 weeks of study product administration.
3. Currently using any medications that may impact dietary fat absorption (i.e., Orlistat, Alli, etc.).
4. Currently using any medications that may interfere with omega-3 uptake (i.e. blood thinning medication or anticoagulants).
5. Currently using any lipid lowering medications (i.e. any cholesterol or triglyceride lowering agent).
6. Currently consuming high amounts of EPA & DHA in the diet (as defined by greater than 200 mg/day by FFQ)
7. Currently following a self-reported no-fat or ultra-restrictive (less than 15%) Low-Fat Diet
8. Having the following medical conditions:

   i. Malabsorptive disorders including but not limited to pancreatitis, Crohn's disease, etc.

   ii. Hypertriglyceridemia (as defined by the Inclusion and per PI discretion; Total cholesterol > 240 mg/dl; LDL > 160 mg/dl; TG > 199 mg/dl) iii. Type2 Diabetes Mellitus
9. Currently a smoker or nicotine user or has been nicotine free for less than 6 months
10. Use of any systemic medications, including OTC medications, herbal products, dietary supplements or vitamins (not previously listed) within 1 week of study product administration (occasional use of OTC analgesics such as acetaminophen may be allowed as judged by the Investigator)
11. Evidence or history of allergic or adverse responses to either study product, any of the product excipients or any comparable or similar products
12. Subjects who are not willing and not able to comply with scheduled visits and the requirements of the study protocol.
13. Female subjects who are breastfeeding, pregnant or plan to become pregnant during this study.
14. Current employee or immediate family member of the study sponsor or study site personnel.
15. Currently participating or have participated in another clinical trial within 4 weeks of study product administration
16. Donated blood, blood components, or significant loss of blood within 30 days of study product administration
17. History of a clinically-significant illness within 4 weeks of study product administration
18. History of hospitalization or treatment for clinically-significant drug or alcohol use/abuse within 1 year of dosing.
19. Subject has poor venous access or difficulty swallowing capsules
20. Any other issue which, in the judgment of the Investigator, will make the subject ineligible for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
AUC0-t | from 0 to 24 hours
  The plasma pharmacokinetics (AUC0-t) resulting from a single oral dose administration will be estimated from 0 to 24 hours post-dose

SECONDARY OUTCOMES:
AUC0-inf | from 0 to infinity
  The plasma pharmacokinetics (AUC0-t) resulting from a single oral dose administration will be estimated from o to infinity
Cmax | between 0 and 24 hours
  The plasma pharmacokinetics (Cmax) resulting from a single oral dose administration will be estimated from 0 to 24 hours post-dose
tmax | between 0 and 24 hours
  The plasma pharmacokinetics (tmax) resulting from a single oral dose administration will be estimated from 0 to 24 hours post-dose
t½ | between 0 and 24 hours
  The plasma pharmacokinetics (t1/2) resulting from a single oral dose administration will be estimated from 0 to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Diane Krieger, MD, Principal Investigator — QPS-MRA
Locations (1):
- QPS/Miami Research Associates, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No